CLINICAL TRIAL: NCT05609994
Title: ViCToRy: Vorasidenib in Combination With Tumor Specific Peptide Vaccine for Recurrent IDH1 Mutant Lower Grade Gliomas
Acronym: ViCToRy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Katy Peters, MD, PhD (Other)
Collaborators: Servier (Industry)
Responsible Party: Sponsor-Investigator, Katy Peters, MD, PhD, Sponsor-Investigator, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00108636
Record Dates: First submitted 2022-11-02; First posted 2022-11-08 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Low Grade Glioma of Brain
Keywords: low grade glioma; brain cancer; vorasidenib; peptide vaccine; immunotherapy; recurrent glioma; Katherine Peters; Pro00108636; IDH mutant
MeSH Terms: conditions — Brain Neoplasms; Glioma | interventions — vorasidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PEPIDH1M vaccine + vorasidenib (Experimental): Patients will receive vaccination with 0.5 mL of Td (tetanus and diphtheria toxoids) intramuscularly into the deltoid muscle. Patients will then receive vorasidenib 40mg orally once a day for 28 days. After two cycles of 28-day vorasidenib and at the start of the 3rd cycle of vorasidenib, patients will receive the PEPIDH1M vaccine intradermally (i.d.) to alternating groin regions on the following schedule: vaccine #1, day 1; vaccine #2, day 15. The day before vaccine #1, patients will receive a vaccine site pre-conditioning injection of a single dose of Td toxoid. This will be administered twelve hours to one day prior to receiving PEPIDH1M vaccine i.d. to the RIGHT groin area. Vaccines #3 and #4 will be given on day 1 and day 15 of cycle 4. Starting on 6th cycle of 28-day vorasidenib, subjects will receive PEPIDH1M vaccine (i.d. to alternating groin regions) every 28 days on day 1 for vaccine #5-#12. Patients will receive up to a total of 14 cycles of vorasidenib.
  Interventions: Drug: PEPIDH1M vaccine + vorasidenib

INTERVENTIONS:
Drug: PEPIDH1M vaccine + vorasidenib — Patients will receive vaccination with 0.5 mL of Td (tetanus and diphtheria toxoids) intramuscularly into the deltoid muscle. Patients will then receive vorasidenib 40mg orally once a day for 28 days. After two cycles of 28-day vorasidenib and at the start of the 3rd cycle of vorasidenib, patients will receive the PEPIDH1M vaccine intradermally (i.d.) to alternating groin regions on the following schedule: vaccine #1, day 1; vaccine #2, day 15. The day before vaccine #1, patients will receive a vaccine site pre-conditioning injection of a single dose of Td toxoid. This will be administered twelve hours to one day prior to receiving PEPIDH1M vaccine i.d. to the RIGHT groin area. Vaccines #3 and #4 will be given on day 1 and day 15 of cycle 4. Starting on 6th cycle of 28-day vorasidenib, subjects will receive PEPIDH1M vaccine (i.d. to alternating groin regions) every 28 days on day 1 for vaccine #5-#12. Patients will receive up to a total of 14 cycles of vorasidenib.

SUMMARY:
The purpose of this study is to determine the safety and efficacy of a PEPIDH1M vaccine in combination with vorasidenib, a dual inhibitor of mutant IDH1 and IDH2 enzymes, in adult patients diagnosed with recurrent IDH1 mutant lower grade gliomas.

DETAILED DESCRIPTION:
This study is designed to assess the safety and efficacy of the PEPIDH1M vaccine in combination with vorasidenib in adult patients recurrent IDH1 mutant lower grade gliomas. Patients will receive vaccination with 0.5 mL of Td (tetanus and diphtheria toxoids adsorbed) intramuscularly (I.M.) into the deltoid muscle to ensure adequate immunity to the tetanus antigen. Patients will then receive vorasidenib 40 mg orally once a day for 28 days. After two cycles of 28-day vorasidenib and at the start of the 3rd cycle of vorasidenib, patients will receive the PEPIDH1M vaccine intradermally (i.d.) to alternating groin regions on the following schedule: vaccine #1, day 1; vaccine #2, day 15. The day before vaccine #1, patients will receive a vaccine site pre-conditioning injection of a single dose of Td toxoid (1 flocculation unit [Lf] in a total volume of 0.4 mL saline). This will be administered twelve hours to one day prior to receiving PEPIDH1M vaccine i.d. to the RIGHT groin area. Vaccines #3 and #4 will be given on day 1 and day 15 of cycle 4. Starting on 6th cycle of 28-day vorasidenib, subjects will receive PEPIDH1M vaccine (i.d. to alternating groin regions) every 28 days on day 1 for vaccine #5-#12. Patients will receive up to a total of 14 cycles of vorasidenib. Notably, a safety lead-in will be performed before commencing on the full study to assess the safety of the combination and evaluation for any dose-limiting toxicity (DLT).

The most common side effects of peptide vaccines are redness or swelling at the injection site, local changes to the texture of skin (hardening) at the injection site, itching, allergic reactions, and a potentially serious side effect called cytokine release syndrome. The most common side effects of vorasidenib are abnormal liver function tests, QT prolongation, stomach and/or intestinal ulcers, neurologic disturbances, skin peeling, and isocitrate dehydrogenase (IDH) differentiation syndrome.

All patients who receive any protocol treatment will be included in either primary or secondary efficacy analyses. Statistical analyses for the primary objective of adverse experience will exclude patients who terminate protocol treatment prematurely (i.e., less than 4 vaccinations) without an unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. IDH1R132H expression in primary tumor
3. Clinical and/or radiographic, progressive Grade 2-3 glioma with greater than 2 cm of non-enhancing disease in one plane.
4. 1st recurrence only
5. Signed informed consent
6. For females of child-bearing potential, negative serum pregnancy test at screening
7. Women of childbearing potential and male participants must agree to practice contraception
8. Karnofsky Performance Status (KPS) of ≥ 70
9. Expected survival of ≥ 12 months
10. Recovered from any clinically relevant toxicities associated with any prior surgery for the treatment of glioma unless stabilized under medical management
11. Complete Blood Count (CBC)/differential with adequate bone marrow function as defined below within 2 weeks of enrollment:

    1. Absolute neutrophil count (ANC) ≥ 1000 cells/mm3
    2. Platelet count ≥ 100,000 cells/mm3
    3. Hemoglobin (Hgb) ≥ 10 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 10 g/dl is acceptable.)
12. Adequate renal function as defined below within 2 weeks of enrollment:

    1. Blood urea nitrogen (BUN) ≤ 25 mg/dl
    2. Creatinine ≤ 1.7 mg/dl
13. Adequate hepatic function as defined below within 2 weeks of enrollment:

    1. Bilirubin ≤ 2.0 mg/dl
    2. Alanine transaminase (ALT) ≤ 3 x normal range
    3. Aspartate aminotransferase (AST) ≤ 3 x normal range

Exclusion Criteria:

1. Prior invasive malignancy (except for non-melanomatous skin cancer) unless disease free for ≥ 3 years (e.g., carcinoma in situ of the breast, oral cavity, and cervix are all permissible)
2. Metastases detected below the tentorium or beyond the cranial vault
3. More than 1 cm X 1 cm of enhancing disease on gadolinium contrasted MRI imaging
4. Severe, active co-morbidity, defined as follows:

   1. Unstable angina and/or congestive heart failure requiring hospitalization
   2. Myocardial infarction within the last 6 months.
   3. Known Acquired Immune Deficiency Syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition (Note: human immunodeficiency virus [HIV] testing is not required for entry into this protocol. The need to exclude patients with Acquired Immunodeficiency Syndrome (AIDS) from this protocol is necessary because treatments involved in this protocol may be significantly immunosuppressive.)
   4. Major medical illnesses or psychiatric impairments that in the investigator's opinion will prevent administration or completion of protocol therapy.
5. Pregnant or lactating women, due to possible adverse effects on the developing fetus or infant due to study drug
6. Patients with a heart-rate corrected QT interval using Fridericia's formula (QTcF) ≥ 450 msec or other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome)
7. Patients with known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection. Subjects with a sustained viral response to HCV treatment or immunity to prior HBV infection will be permitted (Note: Patients with chronic HBV that is adequately suppressed by institutional practice will be permitted.)
8. Patients with active gastrointestinal disease, chronic diarrhea, previous gastric resection or lap band dysphagia, short-gut syndrome, gastroparesis, or other condition that limits the ingestion or gastrointestinal absorption of drugs administered orally (Note: Gastroesophageal reflux disease under medical treatment is allowed.)
9. Patient taking any medications that are CYP3A or CYP2C9 substrates with a narrow therapeutic index (Note: Patients should be transferred to other medications before receiving the first dose of study drug.)
10. Patients treated on any other therapeutic clinical protocols within 30 days prior to study entry or during participation in the study
11. Patients with known hypersensitivity to GM-CSF, yeast-derived products, or any component of Leukine®
12. Allergy or hypersensitivity to tetanus vaccine or any component of the tetanus vaccine.
13. Known hypersensitivity to any component of vorasidenib
14. Prior therapy with mIDH1 targeted therapeutics
15. Unable to undergo MRI imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
To assess the safety of the PEPIDH1M vaccine in combination vorasidenib in adult patients with progressive IDH1 mutant World Health Organization (WHO) Grade 2-3 gliomas | 3.5 years
  The proportion of patients with an unacceptable toxicity
Describe the efficacy, as measured by progression-free survival (PFS), of the combination of PEPIDH1M vaccine and vorasidenib in adult patients with recurrent IDH1 lower grade glioma | 10 years
  The time between initiation of cycle 1 vorasidenib and first documentation of disease progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Peters, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at Duke — http://tischbraintumorcenter.duke.edu/
- See also: Duke Health — http://dukehealth.org/clinical-trials
- See also: Duke Cancer Institute — http://www.dukecancerinstitute.org/